CLINICAL TRIAL: NCT06357650
Title: Protocol for the First Cycle of the Collaborative Open Research Initiative Study (CORIS-1): An International Survey of Personnel in Health Professions Schools
Brief Title: Collaborative Open Research Initiative Study (CORIS-1)
Acronym: CORIS-1
Status: Not yet recruiting | Type: Observational
Sponsor: Chisquares Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: CSQ-2024-001
Record Dates: First submitted 2024-03-20; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Patient Engagement; COVID-19; Preventable Disease, Vaccine; Burnout, Professional; Emerging Infectious Disease; Artificial Intelligence; Climate Change; Online Education; Mental Health Issue; Substance Use Disorders
Keywords: Survey; Global Health; Surveillance; Public health
MeSH Terms: conditions — Patient Participation; COVID-19; Vaccine-Preventable Diseases; Burnout, Professional; Communicable Diseases, Emerging; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Medical schools: Medical schools are institutions offering medical professional degrees like MD, MBBS, or MBChB.
  Interventions: Other: No intervention. This is an observational study
- Dental schools: Dental schools grant dental professional degrees such as DMD, DDS, or BDS.
  Interventions: Other: No intervention. This is an observational study
- Nursing schools: Nursing schools provide degrees or certificates in nursing, including RN and BSc nursing.
  Interventions: Other: No intervention. This is an observational study
- Pharmacy schools: Pharmacy schools offer pharmacy professional degrees, like BPharm or DPharm
  Interventions: Other: No intervention. This is an observational study
- Public health schools: Public health schools encompass programs that confer degrees related to public health practice or research, covering disciplines like epidemiology, biostatistics, health policy, environmental health, ethics, occupational health, global health, and others, including BSc, MPH, DrPH, and MSc.
  Interventions: Other: No intervention. This is an observational study

INTERVENTIONS:
Other: No intervention. This is an observational study — This is an observational study. Hence there is no intervention

SUMMARY:
The Collaborative Open Research Initiative Study (CORIS) is a groundbreaking international research endeavor aimed at exploring vital topics within the field of health professions education. At its core, CORIS embodies the spirit of inclusivity by opening its doors to contributors from all corners of the globe, putting the power of research into the hands of the global community and fostering an environment of open collaboration and meaningful contribution. We invite anyone and everyone to join as collaborators and suggest questions for inclusion in the survey, ensuring that the research process is enriched by diverse perspectives. As a collaborator, you will not only have the opportunity to actively engage in survey design, question formulation, and the entire research process from start to finish, but also gain the prospect of achieving valuable publications, which may boost your professional career.

DETAILED DESCRIPTION:
Introduction:

The Collaborative Open Research Initiative Study (CORIS) embarks on an inclusive and innovative international research endeavor, welcoming contributors from across the globe. CORIS fosters a democratic and collaborative approach, shaping research actively and offering publication opportunities for newcomers in health professions education. We describe CORIS' aims and approach in this study.

Methods:

CORIS, a cross-sectional, web-based survey, seeks to explore critical topics in the field of health professions education. The target population comprises faculty and staff in accredited, degree-granting medical, dental, nursing, pharmacy, and public health schools at both undergraduate and post-graduate levels across 16 countries (n = 14,400). Collaborators can hail from any part of the world but are required to register at https://forms.gle/ZRiwwv3Vmq3y5dv19. Collaborators not only can actively engage in survey design, question formulation, and the entire research process from start to finish but also have the chance to get publications, which can enhance their professional careers. Importantly, there is no financial cost for collaborators at any stage of the study.

Results:

The first iteration, CORIS-1, scheduled for 2024, covers themes such as post-COVID-19 patient care, epidemic preparedness, burnout, artificial intelligence, remote learning, conflict's impact on mental health, substance use, and workplace discrimination. Data will be collected on the Chisquares™ survey platform, and results, codebook, questionnaire, and methods report will be publicly accessible. No sensitive data or identifying information will be collected. CORIS-1 fosters diversity by letting contributors suggest survey questions, aiming to provide novel data, identify gaps, and influence health education policies. It provides an opportunity for research newcomers to engage in the research process from start to finish, and to get publications. Contributors must meet ICMJE authorship criteria. Collaborators can also explore the collected data for their independent projects.

Conclusion:

CORIS redefines research, fostering open collaboration and meaningful contributions. Diverse perspectives and collaborators' contributions are expected to enhance the research process. Graduate students working on theses or dissertations can propose questions in CORIS-1, and early career professionals can also enroll as collaborators to gain a comprehensive understanding of the research process from start to finish.

ELIGIBILITY:
Inclusion Criteria:

The primary data collection targets faculty and staff in accredited, degree-granting medical, dental, nursing, pharmacy, and public health schools, both at the undergraduate and post-graduate levels.

1. Institutional criterion for inclusion is being an accredited program.
2. Individual-level criterion for inclusion is being a faculty or member of staff, including the following categories of personnel: full, associate, and assistant professors; adjunct/part-time/visiting faculty; clinical support staff; research fellows, program coordinators; and administrative staff.

Exclusion Criteria:

1. Residents, teaching assistants, or work-study students who are currently under training.
2. Faculty and staff in post-graduate residency programs that are not degree-awarding.
3. Faculty and staff involved in allied programs, such as dental hygiene, dental assisting, dental technology, pharmacy technology, and medical assistant programs.
4. Faculty members who are either not listed on the online directories of the respective programs or are listed without an email address.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This survey is a cross-sectional, web-based, self-administered questionnaire directed at staff and faculty members in the selected academic programs. We will employ stratified sampling to enhance statistical efficiency, precision, and obtain adequate sample sizes for meaningful inter-group comparisons. The five distinct categories of schools will serve as the strata: (1) Dental schools (2) Medical schools (3) Nursing schools (4) Pharmacy schools (5) Public health schools.
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of health professions schools implementing changes in patient care strategies before versus after the COVID-19 pandemic. | December 2024
  Numerator: Number of individuals within health professions schools who reported a change in patient care strategies due to the COVID-19 pandemic.
  Denominator: Total number of individuals surveyed within health professions schools.
  This indicator assesses the impact of the COVID-19 pandemic on patient care strategies among individuals within health professions schools. It quantifies the proportion of surveyed individuals who have experienced changes in patient care practices, such as telemedicine adoption, virtual consultations, or modifications in clinical rotations, comparing responses collected before and after the onset of the pandemic.
Percentage of personnel in health professions education with adequate epidemic preparedness and readiness. | December 2024
  Numerator: Number of personnel in health professions education who score above a predetermined threshold on the epidemic preparedness and readiness assessment.
  Denominator: Total number of personnel in health professions education assessed for epidemic preparedness and readiness.
Percentage of faculty and staff in health professions schools experiencing burnout. | December 2024
  Numerator: Number of faculty and staff members who meet the criteria for burnout based on standardized assessment tools.
  Denominator: Total number of faculty and staff members surveyed or assessed for burnout.
Percentage of healthcare professionals who report the integration and utilization of artificial intelligence (AI) in their education and practice. | December 2024
  Numerator: Number of healthcare professionals who report using AI in their education and practice.
  Denominator: Total number of healthcare professionals surveyed or assessed for their utilization of AI.
Percentage of participants expressing positive attitudes and perceptions towards climate change and the role of individuals and society in mitigating it. | December 2024
  Numerator: Number of participants expressing positive attitudes and perceptions towards climate change and its mitigation.
  Denominator: Total number of participants surveyed or assessed for their attitudes and perceptions towards climate change.
Percentage of participants reporting effectiveness and challenges of remote learning and online education in health professions schools. | December 2024
  Numerator: Number of participants reporting effectiveness and challenges of remote learning and online education.
  Denominator: Total number of participants surveyed or assessed for their experiences with remote learning and online education in health professions schools.
Percentage of personnel within health professions education reporting substance use behaviors and their implications. | December 2024
  Numerator: Number of personnel reporting substance use behaviors and their implications.
  Denominator: Total number of personnel surveyed or assessed within health professions education.

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study, the data will undergo a thorough cleaning process and be prepared for analysis, alongside the codebook and methodology report which are automatically generated by the Chisquares™ survey platform. All of these materials will be made readily accessible to the public.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: June 1, 2025
Access Criteria: Publicly available to everyone